CLINICAL TRIAL: NCT04590443
Title: Ultrasound-guided Percutaneous Neuromodulation on Hip Muscle Strength
Brief Title: Ultrasound-guided Neuromodulation Percutaneous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Place-NMP
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMP in Infrapiriformis level (Experimental): Participants in this group received NMP of the sciatic nerve in the gluteus region
  Interventions: Other: NMP
- NMP in middle thigh level (Experimental): Participants in this group received NMP of the sciatic nerve in the middle of the thigh
  Interventions: Other: NMP
- NMP in middle distal level (Experimental): Participants in this group received NMP of the sciatic nerve before popliteus region
  Interventions: Other: NMP

INTERVENTIONS:
Other: NMP — Participants received the percutaneous electrical stimulation intervention. Specifically, this consisted of the application of a square wave biphasic electrical current, with 3 Hz frequency and a 250µs pulse width, at the maximal tolerable intensity, to cause an tolerable muscle contraction. The application was 10 stimulations of 10 seconds, with 10 seconds at rest between stimulations. A trained physiotherapist performed the PNM intervention.

SUMMARY:
Chronic low back pain (LBP) is one of the most familiar musculoskeletal pains and alone has been the main origin of years lived with disability for the past three decades. LBP is identified as a nonspecific, painful or mechanical situation in the lower back, buttocks, or hips. Although an underlying origin in chronic LBP has been proposed to be due to a multitude of factors, a muscle hip disbalance has been recognized5. A limited hip internal rotation range of motion (IR-ROM) and hip abductor weakness were found in patients with LBP symptoms7

In the field of Physiotherapy, ultrasound-guided Percutaneous Neuromodulation (PNM) is defined as the application through a needle with ultrasound guidance of an electrical current at low or medium frequency, seeking a sensitive and / or motor response of a peripheral nerve in some point of its trajectory, or of a muscle in a motor point, with a therapeutic objective. However, authors hypothesize that neuromodulation (especially the US-guided PNM technique) may be used to obtain more therapeutic effects, including pain relief.

The main aim of this study was to investigate the effect of hip muscle strengthening by a simple single-shot procedure with the US-guided PNM technique in people with LBP. A second purpose was to discover if the stimulation point in the sciatic nerve territory may influence the change of strength in these patients Sixty subjects will be recruited, which will be divided into 3 groups: group 1 to which PNM will be applied to the sciatic nerve in the gluteus region; group 2 to which PNM will be applied to the sciatic nerve in the middle of the thigh; and group 3 to which PNM will be applied to the sciatic nerve before popliteus region. The PNM intervention with NMP will consist in the single application of an asymmetric rectangular biphasic current (250 microseconds, 3 Hz) during 90 seconds

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lower Back Pain
* Having no other therapy

Exclusion Criteria:

* Other pathology (discal hernia, injured limbs, neurological pathology)
* Belenophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Level of pain | From baseline measurement up to 1 week
  Measured by Visual Analogue Scale (0, no pain; 100, max pain)
Hip internal rotation range of motion | From baseline measurement up to 1 week
  Measured by goniometer.
Muscle strength | From baseline measurement up to 1 week
  Measured by dinamometer. Flexor, extensor, abductor, internal and external rotator muscles
Owestry questionnaire | From baseline measurement up to 1 week
  Lower back pain questionnaire (0, min; 100, max)

CONTACTS AND LOCATIONS:
Locations (1):
- Blanca de la Cruz Torres, Seville, Spain